CLINICAL TRIAL: NCT05570747
Title: Simulated In-House Usability Study of Eclipse Continuous Positive Airway Pressure (CPAP) Device
Status: Completed | Type: Observational
Sponsor: Bleep, LLC (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: BSL-SNAP-001; 1R44HL158286-01A1 (NIH)
Record Dates: First submitted 2022-09-26; First posted 2022-10-07 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — User-Centered Design

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- traditional CPAP Nuance mask users: Human subjects will interact with two different CPAP interfaces including a traditional CPAP mask and the 2nd generation DreamPort-Eclipse. Subjects will be requested to put on each of the different CPAP interface options a total of three times for a total of 6 trials. The order of device tries will be randomized.
  Interventions: Other: Usability
- DreamPort-Eclipse mask users: Human subjects will interact with two different CPAP interfaces including a traditional CPAP mask and the 2nd generation DreamPort-Eclipse. Subjects will be requested to put on each of the different CPAP interface options a total of three times for a total of 6 trials. The order of device tries will be randomized.
  Interventions: Other: Usability

INTERVENTIONS:
Other: Usability — Patients will be observed and asked a serious of questions while they put the mask on and after they remove it.

SUMMARY:
The study is designed to assess the usability of a novel CPAP human interface compared to a traditional nasal mask. Human subjects will interact with two different CPAP interfaces including a traditional CPAP mask and the 2nd generation DreamPort-Eclipse. Subjects will be requested to put on each of the different CPAP interface options a total of three times for a total of 6 trials. The order of device will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years old who are impacted by obstructive sleep apnea and currently are familiar with a CPAP device.

Exclusion Criteria:

* Diagnosis of any medical or behavioral conditions that would compromise subject safety.
* Under the age of 18: target for this current version of the platform is the adult population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were regular clients at the SCMT offices in Murfreesboro and Clarksville. SCMT patients who were already adherent CPAP users were asked if they wanted to participate in research.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Heatherington, Principal Investigator — Bleep, LLC
Locations (3):
- United States (3):
  - AeroFlow Sleep, Asheville, North Carolina
  - Advanced Respiratory and Sleep Medicine, Huntersville, North Carolina
  - Sleep Centers of Middle Tennessee, Murfreesboro, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Data collected through surveys will be available upon request to the principal investigator. Data requested will be de-identified. Only de-identified data will be made available. Only survey responses and the investigators' observational notes, also deidentified, will be shared. No protected health information (PHI) will be shared. Aggregated participant demographic data will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available 4 years after the study completion.
Access Criteria: Requests will be made in writing, to the PI, at stuart@bleepsleep.com. Requests should include the reason for the request, how the data is intended to be used, and additional information may be requested. Data will be shared with credentialed, licensed, or otherwise verifiable researchers/investigators for research purposes only.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study to evaluate the Bleep Eclipse, SCMT patients who were already adherent CPAP users were asked if they wanted to participate in research.
Groups:
- In-House Usability Study Group: Eclipse novel CPAP mask: Participants will follow instructions to set up and put on the Eclipse nasal mask. The Eclipse removes the headgear associated with traditional CPAP masks, offering a small compact design weighing less than an ounce. The Eclipse uses small and lightweight adhesive seals around the nostrils to create an ergonomic design which accommodates the shape of each individual user. It completes a perfect circuit for CPAP therapy to deliver pressure to the airway and stabilize the user's disordered breathing during sleep (apnea and snoring).
  Phillips Respironics Nuance: Participants will follow instructions to set up and put on the Respironics Nuance, traditional nasal mask. Participants will follow instructions to set up and put on the mask. They will fill out a survey about the ease and comfort of putting on and wearing the mask, briefly.
  Participants will follow instructions to set up and put on the mask. They will fill out a survey about the ease and comfort of putting on and wearing the mask, briefly.
Period: Overall Study
Arm/Group | In-House Usability Study Group
Started | 35
Traditional CPAP Mask (Traditional CPAP Mask) | 35 (Each participant wore both the Nuance traditional mask or the Eclipse Novel Mask, in random order, to assess the outcomes. The trials with either mask on, which lasted a few seconds each, were repeated to ensure reproducibility.)
Eclipse Novel CPAP Mask (Experimental mask) | 35 (Each participant wore both the Eclipse Novel Mask or the traditional Nuance mask, in random order, to assess the outcomes. The trials with either mask on, which lasted a few seconds each, were repeated to ensure reproducibility.)
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patient group already being treated at SCMT. Patients were informed about the study and then volunteered to participate if interested.
Groups:
- In-House Usability Study Group: Human subjects will interact with two different CPAP interfaces including a traditional CPAP mask and the 2nd generation DreamPort-Eclipse. Subjects will be requested to put on each of the different CPAP interface options a total of three times for a total of 6 trials. The order of device tries will be randomized.
  Eclipse novel CPAP mask: Participants will follow instructions to set up and put on the Eclipse nasal mask. The Eclipse removes the headgear associated with traditional CPAP masks, offering a small compact design weighing less than an ounce. The Eclipse uses small and lightweight adhesive seals around the nostrils to create an ergonomic design which accommodates the shape of each individual user. It completes a perfect circuit for CPAP therapy to deliver pressure to the airway and stabilize the user's disordered breathing during sleep (apnea and snoring).
  Participants will follow instructions to set up and put on the mask. They will fill out a survey about the ease and comfort of putting on and wearing the mask, briefly.
  Phillips Respironics Nuance: Participants will follow instructions to set up and put on the Respironics Nuance, traditional nasal mask. Participants will follow instructions to set up and put on the mask. They will fill out a survey about the ease and comfort of putting on and wearing the mask, briefly.
Arm/Group | In-House Usability Study Group
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 11
  White | 15
  Hispanic | 6
  Asian | 3

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Each Setup
Description: The estimated time that it takes every subject to place the mask on their faces. Average of 3 trials per mask
Time Frame: Outcomes were assessed on the day of use and only during usage, an average of 20-110 seconds per mask use.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Eclipse Novel CPAP Mask: Human subjects will interact with two different CPAP interfaces including a traditional CPAP mask and the 2nd generation DreamPort-Eclipse. Subjects will be requested to put on each of the different CPAP interface options a total of three times for a total of 6 trials. The order of device tries will be randomized.
  Eclipse novel CPAP mask: Participants will follow instructions to set up and put on the Eclipse nasal mask. The Eclipse removes the headgear associated with traditional CPAP masks, offering a small compact design weighing less than an ounce. The Eclipse uses small and lightweight adhesive seals around the nostrils to create an ergonomic design which accommodates the shape of each individual user. It completes a perfect circuit for CPAP therapy to deliver pressure to the airway and stabilize the user's disordered breathing during sleep (apnea and snoring).
  Participants will follow instructions to set up and put on the mask. They will fill out a survey about the ease and comfort of putting on and wearing the mask, briefly.
- Nuance Traditional Mask: Human subjects will interact with two different CPAP interfaces including a traditional CPAP mask and the 2nd generation DreamPort-Eclipse. Subjects will be requested to put on each of the different CPAP interface options a total of three times for a total of 6 trials. The order of device tries will be randomized.
Arm/Group | Eclipse Novel CPAP Mask | Nuance Traditional Mask
Number analyzed (Participants) | 35 | 35
seconds | 72.9 (26.5) | 14.6 (4.8)

2. Primary Outcome: Number of Technical Issues That Occurred During the Trial
Description: The total number of technical issues that the subject encountered while trying on either mask (average of 3 trials per mask)
Time Frame: Outcomes were assessed on the day of use and only during usage, an average of 20-110 seconds per mask use.
Measure: Mean (Standard Deviation); unit: issues
Arm/Group | Eclipse Novel CPAP Mask | Nuance Traditional Mask
Number analyzed (Participants) | 35 | 35
issues | 6 (1) | 15 (3.4)

3. Primary Outcome: Number of Times Subjects Needed Additional Instructions
Description: The amount of times that the subject needed help from the technician when placing either on either mask. Average of 3 trials per mask.
Time Frame: Outcomes were assessed on the day of use and only during usage, an average of 20-110 seconds per mask use.
Measure: Mean (Standard Deviation); unit: times
Arm/Group | Eclipse Novel CPAP Mask | Nuance Traditional Mask
Number analyzed (Participants) | 35 | 35
times | 3.7 (3.8) | 0 (0)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed on the day of use and only during usage, an average of 20-110 seconds per mask use.
Description: There is some associated risk when completing a clinical trial. The risk for this trial is minimal but is not 0. All 35 participants would have been at risk for a potential adverse event, however, no adverse events were experienced or reported during this study.
Arm/Group | In-House Usability Study Group
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT05570747/Prot_SAP_001.pdf